CLINICAL TRIAL: NCT06801054
Title: Safety Of A Second Dose Of Tenecteplase In Selected Acute Ischemic Stroke Patients Not Responding To The First Dose
Acronym: DoubleDoseTNK
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Hermann Health System (Other)
Collaborators: Grotta Stroke Research Foundation (Unknown); Memorial Hermann Hospital Mobile Stroke Unit (Unknown); The University of Texas Health Science Center, Houston (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, James Grotta, MD, Director Stroke Research and Mobile Stroke Unit, Memorial Hermann Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Double Dose TNK; ML45872 (Other Grant/Funding Number: Houston Mobile Stroke Unit and Genentech)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; tenecteplase; mobile stroke unit; acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tenecteplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving double dose TNK (Experimental): The investigators will give a second dose of IV TNK to patients receiving the initial TNK dose within 3 hrs of LKN, have a baseline NIHSS > 6, and who do not clinically improve within 45 minutes of the first dose, or who improve but then deteriorate, and can still be treated within 4.5 hours from LKN. Patients will require a second CT scan to rule out any bleeding, and meet the usual inclusion and exclusion criteria for TNK treatment, before the second dose which must be given within 4.5 hrs of LKN. Both TNK doses will be 0.25 mg/kg. The initial TNK dose may be given on the MSU or ED, and the second dose in the ED.
  Interventions: Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg)

INTERVENTIONS:
Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg) — All patients will receive a second dose of tenecteplase.

SUMMARY:
In this pilot safety study, the investigators will give a second dose of Intravenous Tenecteplase (IV TNK) to patients receiving the initial TNK dose within 3 hrs of last known normal (LKN), have a baseline National Institutes of Health Stroke Scale (NIHSS) > 6, and who do not clinically improve within 45 minutes of the first dose, or who improve but then deteriorate, and can still be treated within 4.5 hours from LKN. Patients will require a second computed tomography (CT) scan to rule out any bleeding, and meet the usual inclusion and exclusion criteria for TNK treatment, before the second dose which must be given within 4.5 hrs of LKN. Both TNK doses will be 0.25 mg/kg. The initial TNK dose may be given on the Mobile Stroke Unit (MSU) or Emergency Department (ED), and the second dose in the ED. Informed consent will be obtained before the second dose is given.

The primary outcome will be symptomatic intracranial hemorrhage (sICH) (SITS-MOST criteria) or serious systemic bleeding within 36 hours. Secondary outcomes will be any intracranial hemorrhage, any bleeding, discharge NIHSS and modified Rankin Score (mRS), and mRS at 90 days (sliding dichotomy).

20 patients will be enrolled. Enrollment will be stopped if more than 3 sICH occur (> 80% confidence that sICH rate is > 5%. If successful, this study will be followed by a larger phase 2b controlled safety confirmation and pilot efficacy study,

DETAILED DESCRIPTION:
Background: Patients who are eligible for "IVT only" (IVT-O) represent the largest cohort of acute ischemic stroke (AIS) patients who are eligible for IVT, approximately three times larger than those who qualify for both IVT and endovascular thrombectomy (EVT). In all studies of IVT, at least 50% of patients remain disabled at 90 days, generating interest in finding treatments that might augment the beneficial effects of IVT, especially in the majority of AIS patients for whom EVT is not an option. The approved standard doses of tissue plasminogen activator (tPA) and TNK, while based on limited data, suggest that single doses above the approved 0.9 mg/kg of tPA and 0.25 mg/kg TNK will produce excessive bleeding. Another strategy might be to give a second dose of IVT. The relative short half-life of both tPA and TNK after completion of their infusion (5-25 minutes) mean that a second dose might be given while brain tissue is still in the penumbral state which may last for many hours following stroke onset depending on collateral flow. A recent study from France evaluated dual treatment in patients with documented medium vessel occlusion (MeVO) on magnetic resonance angiography (MRA) 1 hour after receiving a single dose of tPA (pts treated within 4.5 hrs of onset and no lesion on magnetic resonance imaging fluid inversion recovery (MRI FLAIR). At one hospital, 146 patients were identified, of whom 96 received TNK on average 116 minutes after tPA. These patients were compared by propensity matching to 148 patients receiving only tPA at another hospital. Dual dose patients showed higher rates of recanalization at 24 hrs (77% vs 61%), better outcome (mRS at 90 days), and no increased bleeding. These very encouraging results in patients limited to those with documented MeVO demonstrate the probable safety of dual IVT dosing and support its ability to increase recanalization in distal vessels thereby improving clinical outcome.

Another strategy would be to use clinical criteria (NIHSS) rather than relying on vascular imaging to identify patients qualifying for a second dose of IVT. The MOST study data demonstrate that 69% of patients with NIHSS > 6 who qualify for IVT and not EVT do not have clot identifiable on vascular imaging and therefore probably harbor more distal occlusions. Furthermore, obtaining a second vascular study 1 hour after the first dose of IVT is problematic at most clinical sites due to lack of availability for obtaining MRA and inability to use CTA due to excessive radiation and contrast. The NIHSS can also be used to identify and exclude those patients who respond to the first dose of IVT. Transcranial doppler studies have shown that early recanalization is associated with rapid clinical improvement on the NIHSS. If the first lytic dose were given within the approved 3 hours, a second dose could still be administered after most of the first dose is dissipated and still within the 4.5 hour time window in those patients who do not clinically improve after the first dose or who initially improve and then deteriorate.

Study Design: In this pilot safety study, the investigators will give a second dose of IV TNK to patients receiving the initial TNK dose within 3 hrs of LKN, have a baseline NIHSS > 6, and who do not clinically improve within 45 minutes of the first dose, or who improve but then deteriorate, and can still be treated within 4.5 hours from LKN. Patients will require a second CT scan to rule out any bleeding, and meet the usual inclusion and exclusion criteria for TNK treatment, before the second dose which must be given within 4.5 hrs of LKN. Both TNK doses will be 0.25 mg/kg. The initial TNK dose may be given on the MSU or ED, and the second dose in the ED. Informed consent will be obtained before the second dose is given.

The primary outcome will be symptomatic ICH (SITS-MOST criteria) or serious systemic bleeding within 36 hours. Secondary outcomes will be any intracranial hemorrhage, any bleeding, discharge NIHSS and mRS, and mRS at 90 days (sliding dichotomy).

20 patients will be enrolled. Enrollment will be stopped if more than 3 sICH occur (> 80% confidence that sICH rate is > 5%. If successful, this study will be followed by a larger phase 2b controlled safety confirmation and pilot efficacy study,

Inclusion criteria for both doses unless indicated otherwise:

* Age 18 and < 80
* Meet standard criteria for TNK
* NIHSS > 6 (for both first and second dose)
* Time from LKN < 3 hrs (first dose) and <4.5 hours (second dose)
* CT at baseline and prior to second dose shows no evidence of intracranial hemorrhage, and ASPECTS > 6.
* No large vessel occlusion (LVO) or EVT
* Pre-stroke mRS < 2

Interventional sequence:

* TNK within 3hr of LKN (all standard criteria met including baseline NIHSS)
* Baseline NIHSS > 6, obtain Informed Consent
* Repeat NIHSS 45 minutes post TNK bolus

  o If repeat NIHSS still > 6, obtain repeat NCCT and review criteria for TNK
* If non contrast CT (NCCT) shows no blood and other criteria for TNK treatment met, give second dose of TNK within 4.5 hrs of LKN (patient enrolled).
* NCCT scan at 24 hrs + 12 or if neurological worsening any time after second dose of TNK
* Neuro checks q 15 min for the first 6 hrs after second dose, then q 60 min for the next 6 hrs
* NIHSS at 24 (+/- 3) hrs from LKN
* NIHSS and mRS at discharge
* mRS at 90 (+/- 14) days from LKN

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms suggestive of acute ischemic stroke
* Age > 18 and < 80 years
* Time from LKN < 3 hrs (first dose) and <4.5 hours (second dose)
* NIHSS > 6 and (for both first and second dose)
* CT at baseline and prior to second dose shows no evidence of intracranial hemorrhage and has an ASPECTS score > 6
* Patient/legally authorized representative has signed the Informed Consent Form

Exclusion Criteria:

* Patients with LVO or MeVO for whom EVT is intended at any time before the second dose of TENECTEPLASE
* At the time of the second dose, NIHSS is < 6
* Systolic blood pressure > 180 at the time of either dose of TENECTEPLASE
* Pre-stroke mRS > 2
* Patients receiving more than one antiplatelet agent during the 48 hours prior to enrollment
* Active internal bleeding
* Patients with undiagnosed significant cognitive impairment or known cerebral amyloid angiopathy
* Patients taking lecanemab, donanemab, or other amyloid reduction therapy
* Known bleeding diathesis
* Recent use of heparin with PTT > control
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; known administration of warfarin within 24 hours or suspected use and INR > 1.5.
* Use of one of the direct oral anticoagulants within the last 48 hours (dabigatran, rivaroxaban, apixaban, edoxaban)
* Treatment with a thrombolytic within the last 3 months prior to enrollment
* Baseline platelet count < 100,000/μL (results must be available prior to treatment)
* Baseline blood glucose > 400 mg/dL (22.20 mmol/L)
* Baseline blood glucose < 50 mg/dL needs to be normalized prior to enrollment
* Intracranial or intraspinal surgery or trauma within 2 months
* History of acute ischemic stroke in the last 90 days
* History of hemorrhagic stroke
* Presumed septic embolus; suspicion of bacterial endocarditis
* Other serious, advanced, or terminal illness (investigator's judgment) or life expectancy is less than 6 months
* Pregnant
* Current participation in another investigational drug or device study
* Known hypersensitivity or allergy to any ingredients of TENECTEPLASE

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients with symptomatic intracerebral hemorrhage or major systemic bleeding | within 36 hours of enrollment (2nd dose of tenecteplase)
  A type 2 parenchymal hemorrhage or a parenchymal hemorrhage remote from the area of infarction with neurological deterioration (≥4-point worsening in National Institutes of Health Stroke Scale) and major hemorrhage (requiring >2 units packed red blood cells)

SECONDARY OUTCOMES:
Clinical efficacy outcome | 90 days post stroke
  National Institutes of Health Stroke Scale (range 0-42 points with lower score indicating less severe stroke) and modified Rankin scale (range 0-6 with lower score indicating less disability)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical and outcome data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after study completion (start date), 5 years after study completion (end date)
Access Criteria: Any academic investigator upon written request to the principal investigator